CLINICAL TRIAL: NCT03994029
Title: The Effects of Polyphenol Supplementation on Hepatic Steatosis, Intima-media Thickness and Non-invasive Vascular Elastography in Obese Adolescents
Brief Title: Effect of Polyphenol Supplementation on Hepatic Steatosis and Vascular Compliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Ramy El Jalbout, Assistant professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-2278
Record Dates: First submitted 2019-06-12; First posted 2019-06-21 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Obesity, Childhood; Hepatic Steatosis; Intimal Hyperplasia
MeSH Terms: conditions — Pediatric Obesity; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyphenol supplementation (Experimental): 120mg per day of powder polyphenol for 60 days
  Interventions: Dietary Supplement: Effect of polyphenols on hepatic steatosis and vascular elastography and intima media thickness
- Placebo (Placebo Comparator): 1 tab PO QD per day of placebo for 60 days
  Interventions: Dietary Supplement: Effect of polyphenols on hepatic steatosis and vascular elastography and intima media thickness

INTERVENTIONS:
Dietary Supplement: Effect of polyphenols on hepatic steatosis and vascular elastography and intima media thickness — Measurement of effect of polyphenol supplementation vs placebo on hepatic steatosis and vascular elastography and intima media thickness

SUMMARY:
The main objective is to study the effect of polyphenol supplementation on hepatic steatosis as measured by hepatic ultrasound, hepatic magnetic resonance imaging and on intima-media thickness and vascular elastography in obese adolescents known for hepatic steatosis as diagnosed by liver biopsy

DETAILED DESCRIPTION:
1. Evaluate the feasibility of a larger, open-label, randomized, controlled trial on the effects of polyphenol supplementation:

   Recruitment, compliance to polyphenol supplementation and the visit roadmaps Duration of the radiological exams and participants' satisfaction and point of view on the experience. Test the relevance of using a food diary. Test the effectiveness of the data collection procedure during the visits. Explore the obstacles encountered while performing the radiological exams and the rate of adverse events (AE). Calculate the sample size of the future randomized clinical study
2. Effects of polyphenols IMT and vascular elastography. Anthropometric measurements, insulin resistance, inflammation, lipid/lipoprotein profile, gut microbiome and liver function
3. Evaluated different imaging modality for steatosis Different imaging modalities will be compared between children

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 18 years
* BMI percentile > 85th for age and sex
* Diagnosis of hepatic steatosis on imaging (ultrasound or MR).
* Diagnosis of hepatic steatosis, NASH, or fibrosis on liver biopsy.
* Elevated alanine aminotransferase (ALT) enzyme level.
* Index of hepatic steatosis 8xALT/AST + BMI (+2 for girls) > 30.

Exclusion Criteria:

* Known chronic systematic diseases
* Any other serious conditions which, according to the doctor's judgment, would prevent compliance and safe participation in the study until completion.

Exclusion criteria to be validated when contacting the participants and their parents/tutors:

* Being pregnant.
* Taking all kinds of prescription or over-the-counter natural health products/natural supplements/vitamins on an ongoing basis or within the next four months, excluding vitamin D.
* Weight loss of 5% to 10% of the usual weight in the last six months before recruitment or weight change of 5% in the last three months.
* Alcohol consumption > two drinks/day or > one day/week.
* Known peanut allergy and/or to the medicinal ingredients contained in the active polyphenol supplement: elderberry, haskap, black chokeberry, blueberry, blackcurrant.
* Any contraindications for MRI.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Through study completion an average of 1 year
  Rate of recruitment
Retention: | Through study completion an average of 1 year
  The percentage of adolescents who agree to participate in the study and the retention
Compliance with polyphenol supplementation | Through study completion an average of 1 year
  Percentage of compliance
Effectiveness of the data collection procedure during the visits | Through study completion an average of 1 year
  Percentage of completed visits
Adverse event | Through study completion an average of 1 year
  Percentage of adverse events
Satisfaction of the participants and their point of view on the experience | Through study completion an average of 1 year
  Percentage of satisfaction of participants enrolled
Sample size calculation for a randomized controlled study | Through study completion an average of 1 year
  A sample size for a future randomized controlled study will be calculated from the estimates obtained during this pilot study.

SECONDARY OUTCOMES:
Change in hepatic steatosis MR | At recruitment, after 60 days, and after 120 days
  mDixonQuant in percentage
Change in hepatic steatosis B-mode US | At recruitment, after 60 days, and after 120 days
  US liver echogenicity normal or increased
Change in intima media thickness (vascular compliance) | At recruitment, after 60 days, and after 120 days
  Measurement of carotid artery intima media thickness in mm
Metabolic syndrome | At recruitment, after 60 days, and after 120 days
  Insulin resistance evaluated by HOMA-IR mg\dl
Cholesterol | At recruitment, after 60 days, and after 120 days
  Triglyceride index (no unit)
Anthropometric measure | At recruitment, after 60 days, and after 120 days
  Body mass index
Inflammatory marker 1 | At recruitment, after 60 days, and after 120 days
  CRP
Inflammatory marker 2 | At recruitment, after 60 days, and after 120 days
  TNF alpha
Inflammatory marker 3 | At recruitment, after 60 days, and after 120 days
  IL-6
Lipid markers 1 | At recruitment, after 60 days, and after 120 days
  Triglycerides
Lipid markers 2 | At recruitment, after 60 days, and after 120 days
  LDL
Lipid markers 3 | At recruitment, after 60 days, and after 120 days
  HDL
Lipid markers 4 | At recruitment, after 60 days, and after 120 days
  Apo AI
Lipid markers 5 | At recruitment, after 60 days, and after 120 days
  Apo B-100
Lipid markers 6 | At recruitment, after 60 days, and after 120 days
  Adiponectin, leptin
Liver function test | At recruitment, after 60 days, and after 120 days
  ALT
Stool test | At recruitment, after 60 days, and after 120 days
  Gut microbiome composition

CONTACTS AND LOCATIONS:
Overall Officials: Ramy El Jalbout, MD MSc, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moretti JB, Drouin A, Truong C, Youn E, Cloutier A, Alvarez F, Paganelli M, Grzywacz K, Jantchou P, Dubois J, Levy E, El Jalbout R. Effects of polyphenol supplementation on hepatic steatosis, intima-media thickness and non-invasive vascular elastography in obese adolescents: a pilot study protocol. BMJ Open. 2024 Jan 30;14(1):e074882. doi: 10.1136/bmjopen-2023-074882. PMID 38296273